CLINICAL TRIAL: NCT03742505
Title: Rapid Normalization of Vitamin D Deficiency in PICU: A Multi-Centre Phase III Double-Blind Randomized Controlled Trial
Brief Title: Rapid Normalization of Vitamin D Deficiency in PICU
Acronym: VITdALIZE-KIDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); EURO-PHARM International Canada, Inc. (Other); Canadian Critical Care Trials Group (Other)
Responsible Party: Principal Investigator, James Dayre McNally, Pediatric Intensivist, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VITdALIZE-KIDS
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Pragmatic, Phase III, multi-centre, double-blinded randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization lists will only be accessible to the Methods Centre at the Ottawa Hospital Research Institute and the research pharmacist(s). The active drug and placebo are identical (e.g. colour, consistency, volume, taste, smell, containers).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D (Experimental): Approximately half of the subjects randomized into VITdALIZE-KIDS will be randomized into the Vitamin D Group and will receive a single dose of cholecalciferol at enrolment.
  Participants may also receive standard vitamin D dosing at the discretion of the care team (e.g. 400-1000 IU/day).
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator): Approximately half of the subjects randomized into VITdALIZE-KIDS will be randomized into the Placebo Group and will receive a single dose of placebo at enrolment.
  Participants may also receive standard vitamin D dosing at the discretion of the care team (e.g. 400-1000 IU/day).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — Single enteral cholecalciferol load at a dose of 10,000 IU/kg (maximum 400,000 IU)
  Arms: Vitamin D
Other: Placebo — Single enteral placebo dose equivalent in volume to the appropriate weight-based dose of cholecalciferol
  Arms: Placebo

SUMMARY:
Vitamin D plays an important role in calcium balance, heart and lung health, inflammation, infection prevention, and muscle strength. Due to these roles, it has been suggested that critically ill patients with low vitamin D levels might have higher rates of death and worse long-term health. We believe that identifying critically ill children with vitamin D deficiency and then restoring vitamin D levels quickly could represent a safe, easy and inexpensive means of reducing patient illness, preventing death and improving quality of life. This clinical trial will determine whether rapid normalization of vitamin D deficiency improves survival and health-related quality of life following critical illness. The VITdALIZE-KIDS trial is a multicentre randomized clinical trial in Canadian Pediatric Intensive Care Units (PICUs). Critically ill children who agree to participate (consent given by caregivers) will have their blood vitamin D level measured, and those who are vitamin D deficient will be randomized to receive a single dose of either high-dose vitamin D3 or placebo (no drug).

Study participants assigned to the high-dose vitamin D arm will receive 10,000 IU/kg of enteral cholecalciferol (up to a maximum of 400,000 IU). We have tested this dose in a pilot trial, and no patient experienced serious adverse events related to vitamin D administration. Patients will be followed for 90 days to determine whether they survived and had a significant change in their health and quality of life. Vitamin D deficiency is a common problem not only among critically ill Canadian children, but in PICUs worldwide. In addition to being applicable in Canada, our study protocol was designed to be generalizable and meaningful to critically ill children worldwide.

DETAILED DESCRIPTION:
Rationale: Documented roles for vitamin D in calcium homeostasis, cardiovascular and respiratory health, innate immunity, and neuromuscular function have led to the hypothesis that vitamin D deficiency (VDD) represents a modifiable risk factor for outcomes in critical illness. Recently, dozens of adult and pediatric intensive care unit (ICU) studies have reported high deficiency rates (50% globally) and associations between VDD, organ dysfunction and mortality. Given the cumulative body of basic science and clinical literature, it has been hypothesized that high-dose vitamin D supplementation could improve ICU outcomes. Recent meta-analyses of multiple small to moderate sized adult clinical trials have suggested improvements in clinical outcome following high-dose supplementation, including survival. Two large multicentre trials have been initiated in the United States and Europe to confirm these findings. In contrast, the benefits and risks of rapid normalization of vitamin D status in the pediatric intensive care unit (PICU) have not been evaluated as part of a large multicentre clinical trial.

Study Design: VITdALIZE-KIDS is a Phase III double blind randomized clinical trial (RCT) to determine whether rapid normalization of VDD in critically ill children improves clinical outcome. In total, 766 critically ill children with VDD will be enrolled from PICUs in Canada.

Objectives: Primary: We will determine if rapid normalization of vitamin D status reduces the decline in health-related quality of life (HRQL), including mortality, that follows pediatric critical illness. Secondary: We will evaluate the impact of rapid normalization of vitamin D status on new or progressive multi-organ dysfunction.

Eligibility Criteria: 1) Admitted to PICU; 2) age 37 weeks corrected gestational age to <18 years; 3) does not meet any exclusion criteria; and 4) blood 25 hydroxyvitamin D (25OHD) under 50 nmol/l. Patients meeting who meet all eligibility criteria and provide consent will be enrolled and randomized.

Interventions: Single dose at enrolment of 10000 IU/kg of cholecalciferol (max 400000 IU) or placebo equivalent in volume to the appropriate dose of cholecalciferol. This dose was evaluated in our pilot dose evaluation trial and shown to be effective (raised group 25OHD levels >75 nmol/L in >75% of participants) and safe (no cases of hypercalcemia or nephrocalcinosis, no difference in the rate of hypercalciuria between study arms). Participants may also receive standard vitamin D dosing at the discretion of the care team (e.g. 400-1000 IU/day).

Data Collection: Baseline HRQL (prior to admission) will be obtained within 72 hours of study enrollment. Follow-up measurements will be obtained in person (for patients who are still in hospital) or by telephone (for patients who have been discharged from hospital) at 28 and 90 days. Data on organ dysfunction, demographics, hospital course, adverse events, and health resource utilization will be collected throughout PICU and hospital stay. A blood sample collected at enrollment on Day 5 (range: Day 3-7) to determine 25OHD response and evaluate vitamin D axis functioning. A urine sample will be collected an enrollment and on Day 5 (range: Day 3-7) for analysis of calcium:creatinine ratio. Sample collection will only be done until 100 patients with full sample collection have been enrolled. Full sample collection is defined as one pre-intervention drug and urine sample and one post-intervention blood and urine sample.

Significance: High VDD rates in PICUs and the recognized interaction between vitamin D status and the health of multiple organ systems suggests vitamin D could represent an inexpensive and safe means of improving outcome. However, the true benefits or risks have not been evaluated in PICU in a clinical trial. The proposed trial seeks to address this question. Study findings will be used to inform guidelines for vitamin D supplementation in PICU, which will be easily generalizable to critically ill children worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to PICU
* Corrected gestational age 37 weeks to age 18 years
* Vitamin D deficiency, as defined by blood 25OHD < 50 nmol/L at the time of screening

Exclusion Criteria:

* Patient will be discharged from PICU before they can be enrolled (i.e. study drug administered) into the VITdALIZE-KIDS study and/or patient will be in hospital for <3 days following enrollment
* Treating physician refuses enteral drug administration due to gastrointestinal disorder, and expects to do so for the full duration of the patient's PICU admission
* Persistent hypercalcemia (ionized calcium >1.40 mmol/L (age >2 months), >1.45 (age <2 months) excluding transient abnormalities and those related to parenteral calcium administration for hypocalcemia;
* Confirmed or suspected William's syndrome;
* Known nephrolithiasis or nephrocalcinosis;
* Imminent plan for withdrawal of treatment or transfer to another ICU not participating in the VITdALIZE-KIDS trial;
* Physician refusal;
* Previous enrollment in this trial;
* Granulomatous disease (tuberculosis or sarcoidosis);
* Severe liver failure;
* Hypersensitivity or allergy to vitamin D or any of the non-medicinal ingredients of the formulation;
* Patient on thiazide diuretics also receiving regular ongoing calcium supplementation above the daily recommended intake;
* Adolescent female of child-bearing age with a positive pregnancy serum test;
* Patient on digoxin-therapy; and
* Treating physician intends to administer vitamin D doses above 1000 IU (e.g. patient presents with isolated clinical symptoms of severe VDD, severe burns).

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 424 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | 28 days
  The primary outcome will be health related quality of life. Health related quality of life will be measures using the age-appropriate PedsQL scale (Ages: 2-7, PedsQL 4.0 Generic Core Scales; Ages 1-24 months: PedsQL™ Infant Core Scales (1-24 months). The PedsQL requires only 23 items to score (36 items for the infant scales), a task easily completed in 5-7 minutes and assesses four domains: physical, emotional, social, and school functioning. The mean PedsQL Core Scale is equal to the sum of all items over the number of items answered on all the Scales and generates a number out of 100. The scoring for the scale is the same for both the PedsQL 4.0 Generic Core Scale and PedsQL Infant Core Scale, allowing the score from either scale to be reported together as one outcome.

SECONDARY OUTCOMES:
New and/or progressive multiple organ dysfunction | 28 days
  The proportion of patients who develop new or progressive multiple organ dysfunction (NPMODS) will be determined using the updated Pediatric Logistic Organ Dysfunction Score (PELOD-2). For patients with no organ dysfunction at randomization, new multiple organ dysfunction syndrome (MODS) will be defined as the development of ≥2 simultaneous organ dysfunctions during the 28 days following randomization (for patients without organ dysfunction at enrolment) or ≥1 simultaneous organ dysfunction (for patients with at least one existing organ dysfunction at enrolment). Progressive MODS will be defined as development of ≥1 additional simultaneous organ dysfunction in a patient with MODS at enrolment. All deaths will be considered Progressive MODS.

OTHER OUTCOMES:
Functional status | 28 and 90 days
  Will be measured using the Functional Status Scale (FSS), which was developed specifically for PICU research, has been both validated against the pediatric performance scales (PCPC/POPC) and has had meaningful change established (3 points). The FSS includes 6 functional domains (mental status, sensory function, communication, motor function, feeding, and respiratory status) and uses a 5-point scale to rate infant function from 1 (normal) to 5 (very severe dysfunction); total scores range from 6 (normal) to 30 (very severe dysfunction).
Mortality | 28 and 90 days
  Consistent with most critical care studies we will evaluate mortality alone
PICU length of stay | Up to 90 days post-randomization
  Duration (in hours and days) of PICU length of stay from time of PICU admission and from time of study enrollment
Hospital length of stay | Up to 90 days post-randomization
  Duration (in days) of hospital length of stay from time of admission and from time of study enrollment
Serious adverse events | Randomization to 90 days post-randomization
  We will report on the frequency of expected and unexpected serious adverse events plausibly associated with vitamin D administration.
Vitamin D toxicity | Randomization to 90 days post-randomization
  We will report on the frequency of biochemical and clinical events potentially related to vitamin-D. Biochemical and clinical events possible related to vitamin D administration include hypercalcemia, nephrocalcinosis/renal stones (symptomatic), and gastric perforation/bleeding.
Change in vitamin D status and axis functioning | Enrolment and on >48 hours following enrollment (range: Day 2-7)
  We will evaluate for change in vitamin D status and axis functioning through blood concentrations of the 1,25(OH)2D and 25OHD metabolites.
Metabolomic profiling | Enrolment and on >48 hours following enrollment (range: Day 2-7)
  Non-targeted metabolomics analysis will be performed on blood and urine using an extensively validated multiplexed separation method for high throughput metabolic phenotyping based on muti-segment injection capillary electrophoresis-mass spectrometry10. This method is applicable to the analysis of a wide array of ionic/polar metabolites in volume-limited biological samples with data fidelity, including matching serum and urine specimens.
Biomarker Analysis - C-Reactive Protein | Enrolment and on >48 hours following enrollment (range: Day 2-7)
  In a sub-set of 100 patients (assuming adequate biological sample volume is obtained), we will report on and compare, by group, the baseline and post-intervention levels of multiple biomarkers shown to be vitamin D responsive in other related populations.
Biomarker Analysis - Pro-inflammatory cytokines | Enrolment and on >48 hours following enrollment (range: Day 2-7)
  In a sub-set of 100 patients (assuming adequate biological sample volume is obtained), we will report on and compare, by group, the baseline and post-intervention levels of multiple biomarkers shown to be vitamin D responsive in other related populations.
Biomarker Analysis - Anti-inflammatory cytokines | Enrolment and on >48 hours following enrollment (range: Day 2-7)
  In a sub-set of 100 patients (assuming adequate biological sample volume is obtained), we will report on and compare, by group, the baseline and post-intervention levels of multiple biomarkers shown to be vitamin D responsive in other related populations.
Biomarker Analysis - Brain natriuretic peptide | Enrolment and on >48 hours following enrollment (range: Day 2-7)
  In a sub-set of 100 patients (assuming adequate biological sample volume is obtained), we will report on and compare, by group, the baseline and post-intervention levels of multiple biomarkers shown to be vitamin D responsive in other related populations.
Biomarker Analysis - Cathelicidin | Enrolment and on >48 hours following enrollment (range: Day 2-7)
  In a sub-set of 100 patients (assuming adequate biological sample volume is obtained), we will report on and compare, by group, the baseline and post-intervention levels of multiple biomarkers shown to be vitamin D responsive in other related populations.
Biomarker Analysis - Bone markers | Enrolment and on >48 hours following enrollment (range: Day 2-7)
  In a sub-set of 100 patients (assuming adequate biological sample volume is obtained), we will report on and compare, by group, the baseline and post-intervention levels of multiple biomarkers shown to be vitamin D responsive in other related populations.

CONTACTS AND LOCATIONS:
Overall Officials: Dayre McNally, MD, PhD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (10):
- Canada (10):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Division of Critical Care, Department of Pediatrics, Victoria Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Centre hospitalier universitaire Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Hearn K, Menon K, Albrecht L, Amrein K, Britz-McKibbin P, Cayouette F, Choong K, Foster JR, Fergusson DA, Floh A, Fontela P, Geier P, Gilfoyle E, Guerra GG, Gunz A, Helmeczi E, Khamessan A, Joffe AR, Lee L, McIntyre L, Murthy S, Parsons SJ, Ramsay T, Ryerson L, Tucci M, McNally D; Canadian Critical Care Trials Group. Rapid normalization of vitamin D deficiency in PICU (VITdALIZE-KIDS): study protocol for a phase III, multicenter randomized controlled trial. Trials. 2024 Sep 19;25(1):619. doi: 10.1186/s13063-024-08461-7. PMID 39300483